CLINICAL TRIAL: NCT04589208
Title: Glutamatergic Mechanisms of Psychosis and Target Engagement (SA1)
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: NIMH institute wide suspension
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Joshua Kantrowitz, Associate Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 8063; R01MH123142-01A1 (NIH)
Record Dates: First submitted 2020-10-13; First posted 2020-10-19 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-07

CONDITIONS: Healthy
Keywords: schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Single blind (rater, participant will be unaware of dose). Subjects will be assigned ketamine doses in 10 subject cohorts
Masking Description: The study will be subject and rater blind, i.e. subjects and raters, will be blinded to the treatment (ketamine dose) group.
  The study physician will be aware of the ketamine dose, and ketamine dose will be the same for both sessions.
  Subjects will not be told what the exact ketamine dose they will receive, but it will be based on their weight and will be no higher than 0.08 mg/kg.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ketamine (Experimental): ketamine
  Interventions: Drug: Ketamine Hydrochloride

INTERVENTIONS:
Drug: Ketamine Hydrochloride — We will assign ketamine doses in successive 10 subject cohorts. The ketamine dose for the 1st cohort will start at 0.08 mg/kg. For subsequent cohorts, the bolus will be successively reduced or increased by 0.02 mg/kg (n=10/dose) to determine the lowest dose of ketamine that still produces a robust phBOLD response

SUMMARY:
50 healthy volunteers (HV) will participate in 2 identical ketamine-induced pharmacoBOLD (phBOLD) sessions at least 7 days apart. On both days, clinical assessments will be performed following removal of the subject from the scanner.

HV will be discharged home after clearance by the study physician. This study will assign ketamine doses in successive 10 subject cohorts. The ketamine dose for the 1st cohort will start at 0.08 mg/kg. For subsequent cohorts, the bolus will be successively reduced or increased by 0.02 mg/kg (n=10/dose) to determine the lowest dose of ketamine that still produces a robust phBOLD response.

The study will be subject and rater blind, i.e. subjects and raters, will be blinded to the treatment (ketamine dose) group.

The study physician will be aware of the ketamine dose, and ketamine dose will be the same for both sessions.

Subjects will not be told what the exact ketamine dose they will receive, but it will be based on their weight and will be no higher than 0.08 mg/kg.

DETAILED DESCRIPTION:
Schizophrenia (Sz) is associated with psychotic symptoms, such as hearing voices and paranoid beliefs that remain partially or fully refractory to standard antipsychotic medications for ~2/3 of patients. Alternative, glutamatergic approaches for treatment development have been proposed but have not yet led to FDA-approved medications. Moreover, several glutamate-targeted medications, such as pomaglumetad (POMA), have failed in pivotal clinical trials despite robust effectiveness in preclinical models. A major barrier to effective glutamatergic treatment development is the absence of validated measures for target engagement that can identify effective compounds and guide dose selection. Target" refers to a factor that an intervention is intended to modify, leading to improvement in symptoms, and target engagement biomarkers are a measure of the ability of the intervention to "engage" the target.

As part of the recently completed NIMH multicenter FAST-PS initiative (IRB protocol 6925 and 7285), we evaluated ketamine-induced pharmacoBOLD (phBOLD) in healthy volunteers (HV) as a potential target engagement biomarker for development of metabotropic glutamate (mGluR2/3) agonists, as a prelude to planned studies in Sz. BOLD imaging indirectly measures brain energy, as a proxy for glutamate target engagement.

The present study will (1) build on these initial positive results to develop phBOLD for use in Sz, (2) optimize ketamine dosing to further increase sensitivity of the phBOLD approach, and (3) explore mechanisms of psychosis. The present study will enable a personalized medicine approach to target engagement and dose evaluation in Sz, while, in parallel, evaluating mechanisms in Sz.

The structure of this grant requires successful completion of Specific Aim (SA) 1 over the first 18 months prior to initiation of SA2 and SA3. We will amend the PSF and consent to include a full description of SA's 2 and 3 prior to its initiation.

In FAST-PS, we selected a high dose of ketamine (0.23 mg/kg) in order to produce robust pharmacological effects. Under SA1, we will titrate this dose downward in HV in order to identify doses that produce reduced psychotomimetic effects, but nevertheless sufficiently robust phBOLD effects.

50 HV will participate in 2 identical phBOLD sessions at least 7 days apart. In total, MRI scans will last approximately 45 minutes, including pre and post ketamine scan. The design is based on our published study(Javitt, Carter et al. 2018). On both days, clinical assessments will be performed following removal of the subject from the scanner.

HV will be discharged home after clearance by the study physician. Although we expect all HV to tolerate ketamine challenge, in the case that a subject does not tolerate it well, we have the capability of admitting a HV subject to an inpatient unit for monitoring and treatment if necessary.

SA1 will assign ketamine doses in successive 10 subject cohorts. The ketamine dose for the 1st cohort will start at 0.08 mg/kg. For subsequent cohorts, the bolus will be successively reduced or increased by 0.02 mg/kg (n=10/dose) to determine the lowest dose of ketamine that still produces a robust phBOLD response.

The study will be subject and rater blind, i.e. subjects and raters, will be blinded to the treatment (ketamine dose) group.

The study physician will be aware of the ketamine dose, and ketamine dose will be the same for both sessions.

Subjects will not be told what the exact ketamine dose they will receive, but it will be based on their weight and will be no higher than 0.08 mg/kg.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-55
2. Medically healthy, as assessed by study physician
3. Capable of understanding the study procedures and able to provide informed consent
4. Eligible men and women must agree to use a reliable method of birth control (for example, use of oral contraceptives or Norplant; a reliable barrier method of birth control diaphragms with contraceptive jelly; cervical caps with contraceptive jelly; condoms with contraceptive foam; intrauterine devices; partner with vasectomy; or abstinence) during the study. Women who are post-menopausal or otherwise not of childbearing potential are also eligible.

Exclusion Criteria:

1. Current or past Axis I psychiatric history (including Substance Use Disorder/Alcohol Use Disorder, with the exception of nicotine use disorder)
2. Positive urine toxicology
3. History of recreational ketamine use, recreational PCP use, or an adverse reaction to ketamine. Subjects who have participated in prior research ketamine studies will be eligible. Subjects can have infusions not more frequently than biweekly, and not more than 1/month on average, therefore subjects entering the study will need to wait one month if they had a single infusion and 6 weeks if they have had two closely spaced infusions.
4. History of first-degree relative with schizophrenia
5. Pregnancy or breast-feeding. This exclusion criterion applies only to females of child-bearing potential (not surgically sterilized and between menarche and 1 year postmenopausal). Must test negative for pregnancy at the time of screening based on a serum pregnancy test.
6. History of violence, including any history of using a gun, knife, or other weapon with intent to harm someone, as well as a more than one physical fight without a weapon after the age of 18 years old (not including fights that happen during sports competition).
7. Presence or positive history of significant medical illness, including renal problems (GFR<60), high blood pressure (defined as systolic blood pressure (SBP) > 140 or diastolic blood pressure (DBP) > 90), low blood pressure (SBP < 100, DBP < 60), orthostatic blood pressure at baseline (change in mean arterial pressure [1/3 systolic + 2/3 diastolic] of > 20%), cardiac illness, or clinically significant abnormal screening labs, as determined by the site physician.
8. Subjects with suicidal ideation with intent or plan (indicated by affirmative answers to items 4 or 5 of the Suicidal Ideation section of the baseline C-SSRS) in the 6 months prior to screening or subjects who represent a significant risk of suicide in the opinion of the investigator.
9. Presence or positive history of neurological illness, including seizures, mental retardation or any other disease/procedure/accident/intervention associated with significant injury to or malfunction of the central nervous system (CNS), or history of significant head injury.
10. Metal implants, pacemaker, other metal (e.g., shrapnel or surgical prostheses) or paramagnetic objects contained within the body which may present a risk to the subject or interfere with the MR scan.
11. Medicinal patch, unless removed prior to the MR scan
12. Claustrophobia
13. Currently taking any psychotropic medication, including antidepressant medications, benzodiazepines, antipsychotic medications, mood stabilizers, anti-epileptic medications, and stimulants. We will exclude any subject who requires treatment with any psychotropic medication from one of these classes.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
PhBOLD | Compare within day changes in phBOLD in response to infusion of ketamine, as measured by resting state fMRI. Calculated by post-pre changes, with higher values indicating higher response. Two scans will be completed, 7 days apart
  Pharmacological Blood-oxygen-level Dependent (phBOLD) Response to ketamine
Brief Psychiatric Rating Scale (BPRS) | Compare within day changes in BPRS in response to infusion of ketamine, as measured by the clinical scale. Calculated by post-pre changes, with higher values indicating higher response. Two scans will be completed, 7 days apart
  Clinical rating scale assessing common psychiatric symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- New York State Psychiatric, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
NIMH Data Archive:
Supporting Information: Study Protocol
Time Frame: after publication
Access Criteria: Qualified reseaerchers
URL: https://nda.nih.gov/